CLINICAL TRIAL: NCT02347150
Title: International Multicenter Study of In-hospital Outcome of Patients After ICU Discharge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Vila Franca de Xira (Other)
Responsible Party: Principal Investigator, João Gonçalves-Pereira, MD, Hospital Vila Franca de Xira
Other Study IDs: HVFX01
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Hospital Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU LOS>24h: 30-110 patients discharged from the ICU

SUMMARY:
Several patients die in the intensive care unit (ICU) due to their acute disease and comorbid conditions. Moreover, after ICU discharge, some ICU survivors still die in the wards.

Previous studies have shown that the clinical condition of the patient at the time of ICU discharge may influence in-hospital prognosis. Non-modifiable factors, such as age and comorbid conditions certainly play a role. But inflammatory status (especially C-reactive protein - CRP), Sequential organ failure score (SOFA) score and Therapeutic intervention scoring system (TISS) 28 score have also been related with the risk of hospital death.

Admission to a high dependency unit may reduce the ICU length of stay (LOS). This strategy may also help to improve prognosis contributing to further stabilize the patient, facilitate his autonomy and the removal of invasive devices. However the benefit of a step-down strategy (from ICU to a high dependency unit) has never been evaluated.

The development of a score to evaluate the risk of patients discharged from the ICU may help to improve the allocation of resources, either to prolong the ICU stay, or admission to a high dependency units or the ward.

DETAILED DESCRIPTION:
Methods Prospective, observational, international, multicentre study to be conducted in 2 countries (Portugal, Brazil). Inclusion criteria: Each centre may include a maximum of 110 consecutive patients discharged from the ICU with length of stay (LOS)>24h during a 6 month period.

Exclusion criteria: Limitation of care decision Primary objective: To determine the impact in hospital mortality and LOS (ICU and hospital) of a step-down strategy, from the ICU to a high dependency unit, before admission to the ward.

Secondary objectives: To develop and validate a score of the risk of death in the hospital after discharge from the ICU

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients discharged from the ICU with LOS>24h

Exclusion Criteria:

* Presence of limitation of care decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients discharge from the ICU with a ICU LOS>24h
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | 6 months
  In hospital mortality after discharge from the ICU

SECONDARY OUTCOMES:
Hospital length of stay | 6 months
  Time between ICU admission and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: João Goncalves-Pereira, MD, Principal Investigator — Hospital Vila Franca de Xira
Locations (3):
- Portugal (3):
  - Hospital Fernando da Fonseca, Amadora
  - Hospital Nélio Mendonça, Funchal
  - Hospital Vila Franca de Xira, Vila Franca de Xira